CLINICAL TRIAL: NCT01096368
Title: Phase III Randomized Trial of Post-Radiation Chemotherapy in Patients With Newly Diagnosed Ependymoma Ages 1 to 21 Years
Brief Title: Maintenance Chemotherapy or Observation Following Induction Chemotherapy and Radiation Therapy in Treating Patients With Newly Diagnosed Ependymoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0831; NCI-2011-02029 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10-01676; COG-ACNS0831; CDR0000668560; ACNS0831 (Other: Children's Oncology Group); ACNS0831 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Results first posted 2023-03-02 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Anaplastic Ependymoma; Brain Ependymoma; Cellular Ependymoma; Clear Cell Ependymoma; Ependymoma; Papillary Ependymoma
MeSH Terms: conditions — Ependymoma | interventions — Radiotherapy, Conformal; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Watchful Waiting; Observation; Cyclophosphamide; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Mesna; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (chemotherapy, observation) (Experimental): Patients with classic histology(WHO Grade II) supratentorial ependymoma who have undergone microscopic gross total resection (GTR1) or achieved CR either after first or second resection or after post-operative induction chemotherapy are assigned to observation. For patients without GTR1, induction chemotherapy is comprised of vincristine intravenously (IV) over 1 minute on days 1 and 8 of cycles 1 and 2, carboplatin IV over 15-60 minutes on day 1 of cycles 1 and 2, and cyclophosphamide IV over 30-60 minutes on days 1-2 of cycle 1 only. Patients also receive etoposide IV over 60-120 minutes on days 1-3 of cycle 2 only. Cycle 1 continues for 3 weeks and cycle 2 continues for 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Etoposide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Mesna; Drug: Vincristine
- Arm II (radiotherapy, chemotherapy) (Experimental): Patients with supratentorial ependymoma (Grade II without GTR1 or Grade III) or any infratentorial ependymoma who have undergone gross or near total resection (GTR or NTR) or achieved CR either after first or second resection or after post-operative induction chemotherapy are randomized to undergo conformal radiotherapy over 6-7 weeks followed by maintenance chemotherapy. Maintenance chemotherapy comprised of vincristine IV on days 1, 8, and 15 of cycles 1-3 only, etoposide IV over 60-120 minutes on days 1-3, cisplatin IV over 1-8 hours on day 1, and cyclophosphamide IV over 30-60 minutes on days 2-3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients without GTR or NTR at enrollment require induction chemotherapy (see Arm I) and possibly second surgery before randomization.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Etoposide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Mesna; Drug: Vincristine
- Arm III (radiotherapy, observation) (Active Comparator): Patients with supratentorial ependymoma (Grade II without GTR1 or ST Grade III) or any infratentorial ependymoma (Grade II or III) who have undergone gross or near total resection or achieved CR either after first or second resection or after post-operative induction chemotherapy are randomized to undergo conformal radiotherapy over 6-7 weeks and then undergo observation. Patients without GTR or NTR at enrollment require induction chemotherapy (see Arm I) and possibly second surgery before randomization.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Other: Clinical Observation; Other: Laboratory Biomarker Analysis
- ARM IV (radiotherapy, chemotherapy) (Active Comparator): Patients with subtotal resection after induction chemotherapy (see Arm I) and second surgery are nonrandomly assigned to Arm II treatment.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Etoposide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Mesna; Drug: Vincristine

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Patients undergo conformal radiotherapy
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
  Arms: ARM IV (radiotherapy, chemotherapy); Arm II (radiotherapy, chemotherapy); Arm III (radiotherapy, observation)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm I (chemotherapy, observation)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: ARM IV (radiotherapy, chemotherapy); Arm II (radiotherapy, chemotherapy)
Other: Clinical Observation — Patients undergo observation
  Other Names: observation
  Arms: Arm III (radiotherapy, observation)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
  Arms: ARM IV (radiotherapy, chemotherapy); Arm I (chemotherapy, observation); Arm II (radiotherapy, chemotherapy)
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP16
  Arms: ARM IV (radiotherapy, chemotherapy); Arm I (chemotherapy, observation); Arm II (radiotherapy, chemotherapy)
Biological: Filgrastim — Given SC or IV
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
  Arms: ARM IV (radiotherapy, chemotherapy); Arm I (chemotherapy, observation); Arm II (radiotherapy, chemotherapy)
Other: Laboratory Biomarker Analysis — Optional correlative studies
Drug: Mesna — Given IV
  Other Names: 2-Mercaptoethanesulfonate, Sodium Salt; Ausobronc; D-7093; Filesna; Mercaptoethane Sulfonate; Mercaptoethanesulfonate; Mesnex; Mesnil; Mesnum; Mexan; Mistabron; Mistabronco; Mitexan; Mucofluid; Mucolene; UCB 3983; Uromitexan; Ziken
  Arms: ARM IV (radiotherapy, chemotherapy); Arm I (chemotherapy, observation); Arm II (radiotherapy, chemotherapy)
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
  Arms: ARM IV (radiotherapy, chemotherapy); Arm I (chemotherapy, observation); Arm II (radiotherapy, chemotherapy)

SUMMARY:
The primary aim of this randomized phase III trial was to study whether the addition of maintenance chemotherapy delivered after surgical resection and focal radiation would be better than surgery and focal radiation alone. The trial also studied if patients who received induction chemotherapy and then either achieved a complete response or went on to have a complete resection would also benefit from maintenance chemotherapy. Children ages 1-21 years with newly diagnosed intracranial ependymoma were included. There were 2 arms that were not randomized. One arm studied patients with Grade II tumors located in the supratentorial compartment that were completely resected. One arm studied patients with residual tumor and those patients all received maintenance chemotherapy after focal radiation. Chemotherapy drugs, such as vincristine sulfate, carboplatin, cyclophosphamide, etoposide, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving chemotherapy in combination with radiation therapy may kill more tumor cells and allow doctors to save the part of the body where the cancer started.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the event free survival (EFS) and overall survival (OS) of children with completely resected ependymoma treated with post-operative conformal radiation therapy (cRT) and then randomized to receive or not receive four cycles of post radiation maintenance chemotherapy (vincristine, cisplatin, etoposide and cyclophosphamide [VCEC]).

EXPLORATORY OBJECTIVES:

I. To estimate the EFS and OS of children with incompletely resected ependymoma who are unable to achieve a complete response (CR) by post-operative induction chemotherapy or by second surgery who will then be non-randomly assigned to cRT followed by four cycles of maintenance chemotherapy (VCEC).

II. To further evaluate the EFS and OS of children with supratentorial classic ependymoma who achieve a complete resection at first or second resection OR children who achieve a CR to short course induction chemotherapy following first surgery.

III. To evaluate whether the addition of maintenance chemotherapy post-radiation therapy contributes to neurobehavioral morbidity and reduced functional outcomes over time, compared to patients treated with radiation therapy followed by observation alone.

IV. To examine differences in neurobehavioral outcomes and quality of life of children treated with proton beam radiation therapy compared to children treated with conventional radiation delivery techniques.

V. To evaluate biologic prognostic factors in childhood ependymoma by studying molecular groups as defined by deoxyribonucleic acid (DNA) methylation profiling and immunohistochemistry, copy number variants to identify 1q gain in posterior fossa ependymomas, CDKN2A loss (homozygous deletion) in supratentorial ependymomas and specific genetic alterations such as RELA fusions, YAP1 fusions and the H3 K27M mutation on initial tumor samples and correlating these data with clinical outcome.

Va. To explore prognostic molecular signatures and genomic alterations in ependymomas by building upon the data derived from ACNS0121 to correlate biomarkers listed above with World Health Organization (WHO) grade, location, extent of resection, treatment, EFS and OS.

OUTLINE: This is a multicenter study partially randomized phase III study. Patients are randomized or non-randomly treated according to tumor location and extent of surgical resection or post-surgery induction chemotherapy response.

Arm I: Patients with classic histology(WHO Grade II) supratentorial ependymoma who have undergone microscopic gross total resection (GTR1) or achieved CR either after first or second resection or after post-operative induction chemotherapy are assigned to observation. For patients without GTR1, induction chemotherapy is comprised of vincristine intravenously (IV) over 1 minute on days 1 and 8 of cycles 1 and 2, carboplatin IV over 15-60 minutes on day 1 of cycles 1 and 2, and cyclophosphamide IV over 30-60 minutes on days 1-2 of cycle 1 only. Patients also receive etoposide IV over 60-120 minutes on days 1-3 of cycle 2 only. Cycle 1 continues for 3 weeks and cycle 2 continues for 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients with supratentorial ependymoma (Grade II without GTR1 or Grade III) or any infratentorial ependymoma who have undergone gross or near total resection (GTR or NTR) or achieved CR either after first or second resection or after post-operative induction chemotherapy are randomized to undergo conformal radiotherapy over 6-7 weeks followed by maintenance chemotherapy. Maintenance chemotherapy comprised of vincristine IV on days 1, 8, and 15 of cycles 1-3 only, etoposide IV over 60-120 minutes on days 1-3, cisplatin IV over 1-8 hours on day 1, and cyclophosphamide IV over 30-60 minutes on days 2-3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients without GTR or NTR at enrollment require induction chemotherapy (see Arm I) and possibly second surgery before randomization.

ARM III: Patients with supratentorial ependymoma (Grade II without GTR1 or ST Grade III) or any infratentorial ependymoma (Grade II or III) who have undergone gross or near total resection or achieved CR either after first or second resection or after post-operative induction chemotherapy are randomized to undergo conformal radiotherapy over 6-7 weeks and then undergo observation. Patients without GTR or NTR at enrollment require induction chemotherapy (see Arm I) and possibly second surgery before randomization.

ARM IV: Patients with subtotal resection after induction chemotherapy (see Arm I) and second surgery are non-randomly assigned to Arm II treatment.

After completion of study therapy, patients are followed up every 4 months for 5 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be newly diagnosed with histologically confirmed intracranial ependymoma; patients with classic ependymoma (WHO II) or anaplastic ependymoma (WHO III) are eligible, as are various subtypes described as clear cell, papillary, cellular or a combination of the above
* There is no minimum performance level; children with ependymoma may suffer neurologic sequelae as a result of their tumor or surgical measures taken to establish a diagnosis and resect the tumor; in the majority of cases, there is neurologic recovery; neurologic recovery is not likely to be impeded by protocol therapy
* REGULATORY: All patients and/or their parents or legal guardians must sign a written informed consent
* REGULATORY: All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with evidence of metastatic disease will be excluded; any evidence of non-contiguous spread beyond the primary site as determined by pre or post-operative magnetic resonance (MR) imaging of brain, pre or post-operative MR imaging of the spine, and post-operative cerebrospinal fluid (CSF) cytology obtained from the lumbar CSF space (the requirement for lumbar CSF examination may be waived if deemed to be medically contraindicated); CSF cytology from a ventriculostomy or permanent ventriculoperitoneal (VP) shunt that reveals the presence of tumor cells is indicative of metastatic disease
* Patients with a diagnosis of spinal cord ependymoma, myxopapillary ependymoma, subependymoma, ependymoblastoma, or mixed glioma are NOT eligible
* No prior treatment other than surgical intervention and corticosteroids; patients are allowed to have had more than one attempt at resection prior to enrollment
* Pregnant female patients are not eligible for this study
* Post-menarchal females may not participate unless a pregnancy test with a negative result has been obtained
* Males and females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Lactating females may not participate unless they have agreed not to breastfeed a child while on this study

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 479 (Actual)
Dates: Start 2010-05-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Smith, Principal Investigator — Children's Oncology Group
Locations (209):
- United States (181):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (11):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Monash Medical Center-Clayton Campus, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Observation: Patients with classic histology (WHO Grade II) supratentorial ependymoma who have undergone microscopic gross total resection (GTR1) or achieved CR either after first or second resection or after post-operative induction chemotherapy are assigned to observation. For patients without GTR1, induction chemotherapy is comprised of vincristine intravenously (IV) over 1 minute on days 1 and 8 of cycles 1 and 2, carboplatin IV over 15-60 minutes on day 1 of cycles 1 and 2, and cyclophosphamide IV over 30-60 minutes on days 1-2 of cycle 1 only. Patients also receive etoposide IV over 60-120 minutes on days 1-3 of cycle 2 only. Cycle 1 continues for 3 weeks and cycle 2 continues for 4 weeks in the absence of disease progression or unacceptable toxicity.
- Arm II: Randomized to Radiation With Maintenance Chemotherapy: Patients with supratentorial ependymoma (Grade II without GTR1 or Grade III) or any infratentorial ependymoma who have undergone gross or near total resection (GTR or NTR) or achieved CR either after first or second resection or after post-operative induction chemotherapy are randomized to undergo conformal radiotherapy over 6-7 weeks followed by maintenance chemotherapy. Maintenance chemotherapy comprised of vincristine IV on days 1, 8, and 15 of cycles 1-3 only, etoposide IV over 60-120 minutes on days 1-3, cisplatin IV over 1-8 hours on day 1, and cyclophosphamide IV over 30-60 minutes on days 2-3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients without GTR or NTR at enrollment require induction chemotherapy (see Arm I) and possibly second surgery before randomization.
- Arm III: Randomized to Radiation Only: Patients with supratentorial ependymoma (Grade II without GTR1 or ST Grade III) or any infratentorial ependymoma (Grade II or III) who have undergone gross or near total resection or achieved CR either after first or second resection or after post-operative induction chemotherapy are randomized to undergo conformal radiotherapy over 6-7 weeks and then undergo observation.
- Arm IV: Nonrandomly Assigned to Arm II Treatment: Patients with subtotal resection after induction chemotherapy (see Arm I) and second surgery are nonrandomly assigned to Arm II treatment.
- Not Ependymoma or Withdrew Before Radiation: Patients with tumor other than ependymoma or withdrew before protocol-specified radiotherapy administered
Period: Overall Study
Arm/Group | Arm I: Observation | Arm II: Randomized to Radiation With Maintenance Chemotherapy | Arm III: Randomized to Radiation Only | Arm IV: Nonrandomly Assigned to Arm II Treatment | Not Ependymoma or Withdrew Before Radiation
Started | 37 | 167 | 163 | 63 | 49
Completed | 37 | 88 | 154 | 39 | 0
Not Completed | 0 | 79 | 9 | 24 | 49
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 13 | 2 | 4 | 6
Not completed — Withdrawal by Subject | 0 | 52 | 0 | 10 | 14
Not completed — Ineligible | 0 | 3 | 2 | 0 | 25
Not completed — Did not start treatment | 0 | 4 | 4 | 0 | 0
Not completed — Progressive disease | 0 | 6 | 0 | 10 | 3
Not completed — Other | 0 | 0 | 1 | 0 | 0
Not completed — Treated with institutional review | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Observation | Arm II: Randomized to Radiation With Maintenance Chemotherapy | Arm III: Randomized to Radiation Only | Arm IV: Nonrandomly Assigned to Arm II Treatment | Not Ependymoma or Withdrew Before Radiation | Total
Number analyzed (Participants) | 37 | 167 | 163 | 63 | 49 | 479
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 164 | 159 | 62 | 48 | 469
  Between 18 and 65 years | 1 | 3 | 4 | 1 | 1 | 10
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 8.8 [1.8 to 19.4] | 4.4 [1.0 to 19.8] | 4.5 [1.0 to 21.0] | 4.2 [1.0 to 18.9] | 7.5 [1.2 to 18.2] | 5.2 [1.0 to 21.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 78 | 68 | 23 | 27 | 214
  Male | 19 | 89 | 95 | 40 | 22 | 265
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 37 | 30 | 11 | 11 | 94
  Not Hispanic or Latino | 29 | 119 | 129 | 47 | 35 | 359
  Unknown or Not Reported | 3 | 11 | 4 | 5 | 3 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 3 | 0 | 1 | 6
  Asian | 1 | 5 | 6 | 4 | 0 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 3 | 1 | 0 | 5
  Black or African American | 6 | 21 | 10 | 6 | 7 | 50
  White | 24 | 113 | 119 | 43 | 30 | 329
  More than one race | 0 | 4 | 1 | 0 | 2 | 7
  Unknown or Not Reported | 5 | 22 | 21 | 9 | 9 | 66
Region of Enrollment [Number; unit: participants]
  United States | 31 | 142 | 132 | 44 | 42 | 391
  Canada | 5 | 17 | 15 | 10 | 3 | 50
  Australia | 0 | 7 | 14 | 8 | 4 | 33
  New Zealand | 1 | 1 | 2 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) in Children Who Have Completely Resected Ependymoma or Achieved CR and Are Treated With Post-radiation Maintenance Chemotherapy or Post-radiation Observation Only
Description: Kaplan-Meier estimates of EFS are calculated from randomization date to first occurrence of disease progression, disease recurrence, second malignant neoplasm, or death from any cause. The comparison between randomized arms (post-radiation maintenance chemotherapy versus post-radiation observation only) is conveyed by the hazard ratio and 90.46% stagewise adjusted Wald confidence interval.
Time Frame: Up to 10 years after enrollment. 5-year estimates of EFS are presented
Population: Eligible, randomized participants (intent-to-treat)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm II: Randomized to Radiation With Maintenance Chemotherapy | Arm III: Randomized to Radiation Only
Number analyzed (Participants) | 164 | 161
percentage of participants | 69.2 [60.8 to 76.2] | 63.7 [55.1 to 71.1]
Statistical Analysis 1: Comparison: Arm II: Randomized to Radiation With Maintenance Chemotherapy vs Arm III: Randomized to Radiation Only; The study was designed to test the superiority of RT+maintenance vs. RT alone as measured by EFS using the hazard ratio via a 1-sided log-rank test. The planned sample size was 160 subjects per arm. 85 EFS events were needed, which were expected after 8 years of accrual and 2 years of follow-up. At 5% type 1 error, the study had 93% power to detect an increase in 2-year EFS from 75% (RT alone) to 87% (RT+maintenance). The design also incorporated interim analyses for futility and efficacy; Test type: Superiority; p = 0.229, Log Rank — P-value is one-sided. After adjusting for interim analyses, the a priori threshold for significance for the final analysis is one-sided alpha=0.031; Hazard Ratio (HR) = 0.866, 90.46% CI 2-sided [0.627 to 1.197] — Hazard ratio is based on hazard of events for Arm II over hazard of events for Arm III. Confidence interval is stage-wise adjusted for multiple interim analyses

2. Primary Outcome: Overall Survival (OS) in Children Who Have Completely Resected Ependymoma or Achieved CR and Are Treated With Post-radiation Maintenance Chemotherapy or Post-radiation Observation Only
Description: Kaplan-Meier estimates of OS are calculated from randomization date to death from any cause. The comparison between randomized arms (post-radiation maintenance chemotherapy versus post-radiation observation only) is conveyed by the hazard ratio and 90.46% stagewise adjusted Wald confidence interval.
Time Frame: Up to 10 years after enrollment. 5-year estimates of OS are presented.
Population: Eligible, randomized participants (intent-to-treat)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm II: Randomized to Radiation With Maintenance Chemotherapy | Arm III: Randomized to Radiation Only
Number analyzed (Participants) | 164 | 161
percentage of participants | 88.3 [81.8 to 92.6] | 86.9 [79.8 to 91.6]
Statistical Analysis 1: Comparison: Arm II: Randomized to Radiation With Maintenance Chemotherapy vs Arm III: Randomized to Radiation Only; It was planned to test the superiority of RT+maintenance vs. RT alone as measured by OS using the hazard ratio via a 1-sided log-rank test using the planned sample size of 160 subjects per arm which was optimized for the EFS outcome. A one-sided significance threshold of 5% was planned for this comparison as well; Test type: Superiority; p = 0.172, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.757, 90.46% CI 2-sided [0.463 to 1.238] — Hazard ratio is based on hazard of death for Arm II over hazard of death for Arm III. Confidence interval is stage-wise adjusted for multiple interim analyses

3. Other Pre Specified Outcome: EFS in Children Who Have Completely Resected Ependymoma at Initial Surgery and Are Treated With Post-radiation Maintenance Chemotherapy or Post-radiation Observation Only
Description: Kaplan-Meier estimates of EFS are calculated from randomization date to first occurrence of disease progression, disease recurrence, second malignant neoplasm, or death from any cause. The comparison between randomized arms (post-radiation maintenance chemotherapy versus post-radiation observation only) for this stratum is conveyed by the hazard ratio and 95% Wald confidence interval.
Time Frame: Up to 10 years after enrollment. 5-year estimates of EFS are presented.
Population: Eligible, randomized participants (intent-to-treat) in stratum 1 (completely resected ependymom at initial surgery)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm II: Randomized to Radiation With Maintenance Chemotherapy in Stratum 1: Patients with supratentorial ependymoma (Grade II without GTR1 or Grade III) or any infratentorial ependymoma who have undergone gross or near total resection (GTR or NTR) after initial surgery (stratum 1) are randomized to undergo conformal radiotherapy over 6-7 weeks followed by maintenance chemotherapy.
- Arm III: Randomized to Radiation Only in Stratum 1: Patients with supratentorial ependymoma (Grade II without GTR1 or ST Grade III) or any infratentorial ependymoma (Grade II or III) who have undergone gross or near total resection after initial surgery (stratum 1) are randomized to undergo conformal radiotherapy over 6-7 weeks and then undergo observation.
Arm/Group | Arm II: Randomized to Radiation With Maintenance Chemotherapy in Stratum 1 | Arm III: Randomized to Radiation Only in Stratum 1
Number analyzed (Participants) | 144 | 142
percentage of participants | 72.7 [63.8 to 79.8] | 62.9 [53.6 to 70.9]
Statistical Analysis 1: Comparison: Arm II: Randomized to Radiation With Maintenance Chemotherapy in Stratum 1 vs Arm III: Randomized to Radiation Only in Stratum 1; In stratum 1, it was also planned to test the superiority of RT+maintenance vs. RT alone as measured by EFS using the hazard ratio via a 2-sided log-rank test. A two-sided significance threshold of 5% was planned for this comparison; Test type: Superiority; p = 0.096, Log Rank — P-value is two-sided and not adjusted for multiple comparisons for this exploratory subgroup comparison; Hazard Ratio (HR) = 0.701, 95% CI 2-sided [0.461 to 1.068] — Hazard ratio is based on hazard of events for Arm II over hazard of events for Arm III

4. Other Pre Specified Outcome: EFS With Incomplete Resection After Initial Surgery, Then Achieved CR After Induction Chemotherapy or GTR/NTR After Second Surgery and Treated With Post-radiation Maintenance Chemotherapy or Post-radiation Observation Only
Description: as for outcome 3
Time Frame: Up to 10 years after enrollment. 5-year estimates of EFS are presented.
Population: Eligible, randomized participants (intent-to-treat) in stratum 2 (completely resected ependymom at initial surgery)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm II: Randomized to Radiation With Maintenance Chemotherapy in Stratum 2: Patients with supratentorial ependymoma (Grade II without GTR1 or Grade III) or any infratentorial ependymoma with incomplete resection after initial surgery and then CR after induction chemotherapy, or patients with GTR/NTR after second surgery (stratum 2) are randomized to undergo conformal radiotherapy over 6-7 weeks followed by maintenance chemotherapy.
- Arm III: Randomized to Radiation Only in Stratum 2: Patients with supratentorial ependymoma (Grade II without GTR1 or ST Grade III) or any infratentorial ependymoma (Grade II or III) with incomplete resection after initial surgery and then CR after induction chemotherapy, or patients with GTR/NTR after second surgery (stratum 2) are randomized to undergo conformal radiotherapy over 6-7 weeks and then undergo observation.
Arm/Group | Arm II: Randomized to Radiation With Maintenance Chemotherapy in Stratum 2 | Arm III: Randomized to Radiation Only in Stratum 2
Number analyzed (Participants) | 20 | 19
percentage of participants | 41.7 [17.9 to 64.0] | 67.5 [41.4 to 84.0]
Statistical Analysis 1: Comparison: Arm II: Randomized to Radiation With Maintenance Chemotherapy in Stratum 2 vs Arm III: Randomized to Radiation Only in Stratum 2; In stratum 2, it was also planned to test the superiority of RT+maintenance vs. RT alone as measured by EFS using the hazard ratio via a 2-sided log-rank test. A two-sided significance threshold of 5% was planned for this comparison; Test type: Superiority; p = 0.041, Log Rank — P-value is two-sided and not adjusted for multiple comparisons for this exploratory subgroup comparison; Hazard Ratio (HR) = 2.684, 95% CI 2-sided [1.004 to 7.175] — Hazard ratio is based on hazard of events for Arm II over hazard of events for Arm III

5. Other Pre Specified Outcome: OS in Children Who Have Completely Resected Ependymoma at Initial Surgery and Are Treated With Post-radiation Maintenance Chemotherapy or Post-radiation Observation Only.
Description: Kaplan-Meier estimates of OS are calculated from randomization date to death from any cause. The comparison between randomized arms (post-radiation maintenance chemotherapy versus post-radiation observation only) for this stratum is conveyed by the hazard ratio and 95% Wald confidence interval.
Time Frame: Up to 10 years after enrollment. 5-year estimates of OS are presented.
Population: Eligible, randomized participants (intent-to-treat) in stratum 1 (completely resected ependymom at initial surgery)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm II: Randomized to Radiation With Maintenance Chemotherapy in Stratum 1 | Arm III: Randomized to Radiation Only in Stratum 1
Number analyzed (Participants) | 144 | 142
percentage of participants | 90.7 [84.2 to 94.7] | 86.4 [78.5 to 91.5]
Statistical Analysis 1: Comparison: Arm II: Randomized to Radiation With Maintenance Chemotherapy in Stratum 1 vs Arm III: Randomized to Radiation Only in Stratum 1; In stratum 1, it was also planned to test the superiority of RT+maintenance vs. RT alone as measured by OS using the hazard ratio via a 2-sided log-rank test. A two-sided significance threshold of 5% was planned for this comparison; Test type: Superiority; p = 0.067, Log Rank — P-value is two-sided and not adjusted for multiple comparisons for this exploratory subgroup comparison; Hazard Ratio (HR) = 0.547, 95% CI 2-sided [0.284 to 1.053] — Hazard ratio is based on hazard of death for Arm II over death of events for Arm III

6. Other Pre Specified Outcome: OS in Children With Incomplete Resection After Initial Surgery Who Then Achieved CR After Induction Chemotherapy or GTR/NTR After Second Surgery and Are Treated With Post-radiation Maintenance Chemotherapy or Post-radiation Observation Only
Description: as for outcome 5
Time Frame: Up to 10 years after enrollment. 5-year estimates of OS are presented.
Population: Eligible, randomized participants (intent-to-treat) in stratum 2 (induction chemotherapy or second surgery required)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm II: Randomized to Radiation With Maintenance Chemotherapy in Stratum 2 | Arm III: Randomized to Radiation Only in Stratum 2
Number analyzed (Participants) | 20 | 19
percentage of participants | 69.2 [40.2 to 86.2] | 89.5 [64.1 to 97.3]
Statistical Analysis 1: Comparison: Arm II: Randomized to Radiation With Maintenance Chemotherapy in Stratum 2 vs Arm III: Randomized to Radiation Only in Stratum 2; In stratum 2, it was also planned to test the superiority of RT+maintenance vs. RT alone as measured by OS using the hazard ratio via a 2-sided log-rank test. A two-sided significance threshold of 5% was planned for this comparison; Test type: Superiority; p = 0.094, Log Rank — P-value is two-sided and not adjusted for multiple comparisons for this exploratory subgroup comparison; Hazard Ratio (HR) = 3.601, 95% CI 2-sided [0.724 to 17.902] — Hazard ratio is based on hazard of death for Arm II over hazard of death for Arm III

7. Other Pre Specified Outcome: EFS of Children With Incompletely Resected Ependymoma Who Are Unable to Achieve a Complete Response (CR) by Post-operative Induction Chemotherapy or by Second Surgery and Who Are Non-randomly Assigned to Receive Maintenance Chemotherapy
Description: The Kaplan-Meier estimate of EFS is calculated from enrollment date to first occurrence of disease progression, disease recurrence, second malignant neoplasm, or death from any cause.
Time Frame: Up to 10 years after enrollment. 5-year estimates of EFS are presented.
Population: Eligible participants in Arm IV (intent-to-treat)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm IV: Nonrandomly Assigned to Arm II Treatment: Patients with subtotal resection after induction chemotherapy (see Arm I) and second surgery are non-randomly assigned to Arm II treatment.
Arm/Group | Arm IV: Nonrandomly Assigned to Arm II Treatment
Number analyzed (Participants) | 63
percentage of participants | 33.6 [22.1 to 45.5]

8. Other Pre Specified Outcome: OS of Children With Incompletely Resected Ependymoma Who Are Unable to Achieve a Complete Response (CR) by Post-operative Induction Chemotherapy or by Second Surgery and Who Are Non-randomly Assigned to Receive Maintenance Chemotherapy
Description: The Kaplan-Meier estimate of OS is calculated from enrollment date to death from any cause.
Time Frame: Up to 10 years after enrollment. 5-year estimates of OS are presented.
Population: Eligible participants in Arm IV (intent-to-treat)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm IV: Nonrandomly Assigned to Arm II Treatment
Number analyzed (Participants) | 63
percentage of participants | 74.0 [60.5 to 83.5]

9. Other Pre Specified Outcome: EFS of Children With Supratentorial Classic Ependymoma Who Achieve Complete Resection at First or Second Surgery or Children Who Achieve Complete Response (CR) After Induction Chemo and Who Are Non-randomly Assigned to Observation
Description: as for outcome 7
Time Frame: Up to 10 years after enrollment. 5-year estimates of EFS are presented.
Population: Eligible participants in Arm I
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I: Observation
Number analyzed (Participants) | 37
percentage of participants | 66.9 [49.0 to 79.7]

10. Other Pre Specified Outcome: OS of Children With Supratentorial Classic Ependymoma Who Achieve Complete Resection at First or Second Surgery or Children Who Achieve Complete Response (CR) After Induction Chemo and Who Are Non-randomly Assigned to Observation
Description: The Kaplan-Meier estimate of OS is calculated from enrollment date to death from any cause.
Time Frame: Up to 10 years after enrollment. 5-year estimates of OS are presented.
Population: Eligible participants in Arm I
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I: Observation
Number analyzed (Participants) | 37
percentage of participants | 100 [87.2 to 100.0]

ADVERSE EVENTS:
Time Frame: Enrollment up to 10 years after enrollment.
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Arm I: Observation | Arm II: Randomized to Radiation With Maintenance Chemotherapy | Arm III: Randomized to Radiation Only | Arm IV: Nonrandomly Assigned to Arm II Treatment | Not Ependymoma or Withdrew Before Radiation
All-Cause Mortality (participants affected / at risk) | 0/37 | 20/164 | 27/161 | 22/63 | 4/24
Serious Adverse Events (participants affected / at risk) | 0/37 | 5/164 | 0/161 | 1/63 | 0/24
Other Adverse Events (participants affected / at risk) | 0/37 | 22/164 | 10/161 | 15/63 | 4/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Observation (N=37) | Arm II: Randomized to Radiation With Maintenance Chemotherapy (N=164) | Arm III: Randomized to Radiation Only (N=161) | Arm IV: Nonrandomly Assigned to Arm II Treatment (N=63) | Not Ependymoma or Withdrew Before Radiation (N=24)
Death NOS (General disorders) | 0 | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Observation (N=37) | Arm II: Randomized to Radiation With Maintenance Chemotherapy (N=164) | Arm III: Randomized to Radiation Only (N=161) | Arm IV: Nonrandomly Assigned to Arm II Treatment (N=63) | Not Ependymoma or Withdrew Before Radiation (N=24)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 4 | 2 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 6 | 2 | 3 | 1
Platelet count decreased (Investigations) | 0 | 3 | 0 | 3 | 0
White blood cell decreased (Investigations) | 0 | 4 | 2 | 4 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 2 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 3 | 0
Central nervous system necrosis (Nervous system disorders) | 0 | 3 | 3 | 0 | 0
Edema cerebral (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Vagus nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT01096368/Prot_SAP_000.pdf